CLINICAL TRIAL: NCT05167955
Title: A Preliminary Randomised Controlled Study Online Mindfulness-Based-Cognitive-Intervention for African Caribbean Men
Brief Title: Mindfulness-Based-Cognitive-Intervention for African Caribbean Men With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Principal Investigator, London Metropolitan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LondonMU
Record Dates: First submitted 2021-11-19; First posted 2021-12-22 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Erectile Dysfunction
Keywords: sexual wellbeing; mindfulness; sexual self-efficacy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled waitlist (N= 34 experimental and n=34 waitlist)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Randomized controlled waitlist (Experimental): n=34 (will receive Mindfulness-based cognitive intervention)
  Interventions: Behavioral: Mindfulness based cognitive intervention based on the behavioural change techniques taxonomy
- Waitlist Randomized controlled waitlist (Other): waitlist Randomized controlled waitlist n=34 (will not receive Mindfulness-based cognitive intervention for 1 month)
  Interventions: Behavioral: Mindfulness based cognitive intervention based on the behavioural change techniques taxonomy

INTERVENTIONS:
Behavioral: Mindfulness based cognitive intervention based on the behavioural change techniques taxonomy — An online mindfulness-based cognitive intervention is used as a proposed treatment intervention for erectile dysfunction among African- Caribbean men based in the United Kingdom.

SUMMARY:
Title of research: A preliminary Randomised Controlled Study online Mindfulness-Based-Intervention for African-Caribbean men with Erectile Dysfunction

Research aim: How an online mindfulness intervention, based on a behavioral health taxonomy, might reduce symptoms of erectile dysfunction and increase sexual well-being among African-Caribbean men in the United Kingdom.

Research intention: If the Mindfulness-based intervention reduces symptoms of erectile dysfunction and increases sexual wellness, then we would repeat this study on a larger scale among Black, Asian, Minority, and Ethnic men via the National Health Service.

A brief overview of intervention: Erectile dysfunction is the inability to achieve or maintain an erection in up to 75 to 100% of sexual attempts, including masturbation and sexual intercourse. It is typically very costly to treat on the National Health Service, using the combination of medication (e.g. Viagra) and psychosexual therapy.

The use of mindfulness in healthcare for varied psychosocial difficulties is gaining popularity. A meta-analysis on mindfulness and sexual dysfunction among men and women. Whilst gender differences were the priority focus of the analysis, it also looked at how well-represented cultural and minority groups were within the existing clinical trials. The review identified no studies relating to Black, Asian, Minority and Ethnic men with erectile dysfunction and mindfulness.

Quantitatively, the research is structured so that participants will be randomized to either the experimental or control group (n=34 experimental; n=34 control waitlist). A 2-month follow-up will be taken to determine the sustainability of this intervention.

DETAILED DESCRIPTION:
The principal researcher developed the online mindfulness cognitive intervention. An understanding of the intervention along with educational sessions about erectile dysfunction will be carried out among the team. Part of this programme will involve the research assistants who will overview the implementation of the assessments and pre and post output measurements of the intervention. The mindfulness box will include an array of educational material and cognitive templates on erectile dysfunction and sexual behaviour education. The mindfulness specialist will deliver the intervention. In total, 16 domains have been included in the development of this intervention. Of these, 35 out of the 93 behavioral change techniques taxonomy were identified.

The main targets here are to engage those with mindfulness exercises whilst improving wellbeing and minimizing erectile dysfunction. This will aim to show salience of consequences where feedback will emphasize the positive outcomes of performing the mindfulness-based cognitive intervention. The main exercises include mindfulness, breathing exercises, relaxation techniques, being mindful of the senses and the body, and understanding of the self. Each of the 4 sessions will be between 2-3 hours long where at-home exercises will be encouraged.. Feedback and support along with discussing the educational components, training, modelling and enablement will be addressed throughout. As the content of the randomized controlled study online mindfulness-based cognitive intervention is, the specific intervention targets described in table 1 have included cognitive, emotional, or behavioral factors or a combination of these.

Table 1

Techniques within this Intervention target Behaviour change techniques taxonomy Randomised controlled study

Cognitive

Psychoeducation Understanding erectile dysfunction 4.2, 5.1, 5.3, 5.5, 5.6, 9.2 The hot cross bun

Sexual self-efficacy Enjoyable sex 1.2,1.4, 1.9, 2.3, 11.2, 15.3,16.2

Cognitive reframe/self talk Challenging thoughts associated 4.3, 11.2, 13.2, 15.4 with sexual performance

Behavioural

Reward and reinforcement Encourage new behaviour coupled 1.2, 1.4, 4.1, 8.1, 8.2 with positive feedback 10.7, 10.10, 11.2, 14.4

Self-care Behaviours which promote physical 10.7, 10.10 mental and emotional well-being

Self-monitoring Monitor behaviour towards goals 1.1, 1.2, 1.3, 1.4, 1.9, 2.2, 2.3, 2.7

Mindfulness-based cognitive intervention

Understanding emotions Recognising and developing emotions 1.2, 3.1, 5.6, 8.1, 11.2 and coping strategies 12.4

Goal setting/smart goals Specific, Measurable, Achievable, 1.1, 1.2, 1.3, 1.4, 1.9, 2.2,2.3,2.7 Realistic and anchored within a Time Frame.

Self-directed meditation Creating better awareness of 1.9, 4.1, 6.1,8.1, 11.2,15.2 body, mind and breathing

Body scan Bringing attention and awareness 4.1, 6.1, 8.1, 11.2, 15.2 to different areas of the body. Top to toe.

Mindfulness practices Being aware of the present moment 4.1, 6.1,8.1, 11.2, 12.6 15.2, 16.2

Mindfulness stretching Mind and body connection 4.1, 6.1, 8.1, 11.2, 12.6, 15.2, 16.2

Self-compassion Encouraging a positive self-identity 11.2, 13.1, 13.2, 13.4, 13.5

ELIGIBILITY:
Inclusion Criteria:

* African Caribbean men with erectile dysfunction
* Aged 18 years and above
* Registered with a general practitioner

Exclusion Criteria:

* Taking Viagra during the study
* Aged younger than 18 years
* Non-African-Caribbean
* Not registered with a general practitioner

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — African Caribbean men aged 18 years and above with erectile dysfunction
Enrollment: 68 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline in erectile dysfunction on a 5 item questionnaire at 0,4 and 8 weeks | 0 baseline 4, and 8 week measurements
  This consists of 5 questions with 5 response categories measuring erectile functioning, satisfaction and desire for the last 4 weeks. Cronbach alpha= 0.82 to 0.93. The response categories range from 0=no sexual activity to 5=almost always/always. Subscale scoring is divided into 5 areas including sexual activity, sexual intercourse, sexual stimulation, sexual, ejaculation and orgasm. There is no reverse scoring where scores range from 0 to 75, the latter being higher levels of erectile functioning.
Change in baseline in mindfulness on a 10 item questionnaire at 0, 4,and 8 weeks | 0 baseline 4, and 8 week measurements
  This is a 10-item questionnaire which consists of 5 response categories (1=never or rarely true through to 5= very often/always true). Cronbach's alpha ranges between 0.69-0.76. There are 7 reversed items. Subscale scoring is divided into 5 areas including observing, describing, acting with awareness, non-judging and non-reactivity. Higher scores reflect higher levels of mindfulness endorsement.
Change in baseline in wellbeing on a 7 item questionnaire at 0. 4 and 8 weeks | 0 baseline, 4, and 8 week measurements
  A positively worded 7 item questionnaire with 5 response categories looking at functioning and feeling aspects of well-being. The response categories include 1=none of the time to 5=all of the time. Cronbach alpha- 0.89-0.91. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing.
Change in baseline in sexual self-efficacy on a 25 item questionnaire at 0, 4, and 8 weeks | 0 baseline, 4,and 8 week measurements
  The Sexual Self-Efficacy Erectile tool is a 25-item questionnaire which focuses on sexual confidence and behaviour change associated with therapy. Participants responses are measured via a 10-item scale ranging from 10 to 100. Here, 10 is the lowest level of self-efficacy and 100 is the highest. There are no reverse questions. The Cronbach's alpha for men with erectile difficulties is α =0.88 (high) and for men without erectile difficulties, α =0.62 (low to moderate).

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, PhD, Principal Investigator — Reader
Locations (1):
- London Met university, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders: DSM-5. Washington DC: Author.
- [Background] Banbury, S., Lusher, J., Snuggs, S & Chandler, C., (2021). Mindfulness-based therapies for men and women with sexual dysfunction: a systematic review and meta-analysis, Sexual and Relationship Therapy, DOI: 10.1080/14681994.2021.1883578
- [Background] Bossio JA, Basson R, Driscoll M, Correia S, Brotto LA. Mindfulness-Based Group Therapy for Men With Situational Erectile Dysfunction: A Mixed-Methods Feasibility Analysis and Pilot Study. J Sex Med. 2018 Oct;15(10):1478-1490. doi: 10.1016/j.jsxm.2018.08.013. PMID 30297094
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Libman E, Rothenberg I, Fichten CS, Amsel R. The SSES-E: a measure of sexual self-efficacy in erectile functioning. J Sex Marital Ther. 1985 Winter;11(4):233-47. doi: 10.1080/00926238508405450. PMID 4078907
- [Background] Rhoden EL, Teloken C, Sogari PR, Vargas Souto CA. The use of the simplified International Index of Erectile Function (IIEF-5) as a diagnostic tool to study the prevalence of erectile dysfunction. Int J Impot Res. 2002 Aug;14(4):245-50. doi: 10.1038/sj.ijir.3900859. PMID 12152112
- [Background] Feldman, G., Hayes, A., Kumar, S., Greeson, J., & Laurenceau, J. P. (2007). Mindfulness and emotion regulation: The development and initial validation of the Cognitive and Affective Mindfulness Scale Revised (CAMS-R). Journal of Psychopathology and Behavioral Assessment, 29(3), 177-190.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT05167955/Prot_SAP_ICF_001.pdf